CLINICAL TRIAL: NCT04065308
Title: A Phase II Trial to Evaluate the Efficacy of Daratumumab With DCEP in Multiply Myeloma Patients With Plasmacytoma Who Fail to Achieve Complete Remission With Bortezomib Containing Induction Regimen
Brief Title: Daratumumab With DCEP for Multiple Myeloma With Plasmacytoma
Acronym: Dara_DCEP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Youngil Koh, Assistant Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1803-019-927
Record Dates: First submitted 2019-08-21; First posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Multiple Myeloma in Relapse; Plasmacytoma; Daratumumab
MeSH Terms: conditions — Plasmacytoma | interventions — Drug Combinations; daratumumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental arm (Experimental): Daratumumab plus DCEP,combination therapy is administered total of three cycles,every 4weeks(28 days).
  Daratumuamb 16mg/kg body weight in 500mL (the first dose,16mg/kg body weight in 1000mL) Weeks 1 to 8: weekly Weeks 9-24 : every 2 weeks if ASCT ineligible or PR but Plasmacytoma response <CR: every 2 weeks for 12weeks and then every 4 weeks for 8weeks (Total of 8 times, additional administration of daratumumab) if ASCT eligible: From 6 to 12 weeks after ASCT, administration of daratumumab is initiated within 12 weeks of ASCT and twice a month for 12 weeks and then every a months for 8 weeks. (Total of 8 additional administration of daratumumab after ASCT)
  1. dexamethasone :40mg/day D1-4, intravenous
  2. cyclophosphamide: 400mg/m2 D1-4, intravenous
  3. etoposide: 40mg/m2 D1-4, intravenous
  4. cisplatin : 7mg/m2 D1-4, intravenous Pegteograstim: 6mg once, SC on day 5 or 6 of each 28-day cycle
  Interventions: Drug: Drug Combinations

INTERVENTIONS:
Drug: Drug Combinations — Daratumumab plus DCEP,combination therapy is administered total of three cycles,every 4weeks(28 days).
  Daratumuamb 16mg/kg body weight in 500mL (the first dose,16mg/kg body weight in 1000mL) Weeks 1 to 8: weekly Weeks 9-24 : every 2 weeks if ASCT ineligible or PR but Plasmacytoma response <CR: every 2 weeks for 12weeks and then every 4 weeks for 8weeks (Total of 8 times, additional administration of daratumumab) if ASCT eligible: From 6 to 12 weeks after ASCT, administration of daratumumab is initiated within 12 weeks of ASCT and twice a month for 12 weeks and then every a months for 8 weeks. (Total of 8 additional administration of daratumumab after ASCT)
  1. dexamethasone :40mg/day D1-4, intravenous
  2. cyclophosphamide: 400mg/m2 D1-4, intravenous
  3. etoposide: 40mg/m2 D1-4, intravenous
  4. cisplatin : 7mg/m2 D1-4, intravenous Pegteograstim: 6mg once, SC on day 5 or 6 of each 28-day cycle
  Other Names: Daratumumab plus DCEP

SUMMARY:
This trial aimed to investigate the therapeutic efficacy of daratumumnab plus chemitherapy in multiple myeloma with plasmacytoma.

DETAILED DESCRIPTION:
Multiple myeloma with plasmacytoma is a disease with significantly short overall survival. Cancer cells in plasmacytoma has inferior response compared to cancer cells in bone marrow in multiple myeloma. It is revealed that genetic difference such as CCND1 overexpression and RAS mutation exists between plasmacytoma and intramedullary plasma cell myeloma, implying different treatment strategy should be applied to overcome poor prognosis of this distinct disorder.

Even in the era of potent IMiDs and proteasome inhibitors, median overall survival of multiple myeloma patients with plasmacytoma is less than 5 years. Moreover, relapse in a form of soft tissue plasmacytoma is frequently observed after triplet combination treatment in multiple myeloma. Hence, multiple myeloma with plasmacytoma is a disease where unmet medical need still exists.

Biologically, plasmacytoma is characterized by high plasma cell proliferation, angiogenesis gene profile, and adhesion molecule changes mimicking solid tumor . Responsiveness to chemotherapy used in myeloma including IMIds5 and proteasome inhibitor6 is obtuse in plasmacytoma. Only small fraction of young patients receiving high-dose chemotherapy followed by autologous stem cell transplantation may overcome adverse prognostic impact of plasmacytomas . Even it is recommended that VTD-PACE would be used as the first line treatment for plasmacytomas.

In summary, cancer cells in plasmacytoma bear biologic characteristics of solid tumor cells and do respond to high-dose chemotherapy. And this phenomenon is very similar to lymphoma for the following reasons. Like lymphoma, 1) plasmacytoma express tumor antigen strongly (CD38 or CD138), 2) they form a solid mass, and 3) respond to cytotoxic chemotherapy in a dose-response manner.

Considering the success story of rituximab in lymphoma, we conjecture that daratumumab may work excellently to control plasmacytoma. Hence, we propose a treatment regimen consists of DCEP chemotherapy and daratumumab.

ELIGIBILITY:
Inclusion Criteria:

ECOG performance status 2 or better Adequate physical condition that could tolerate cytotoxic chemotherapy judged by investigator Relapsed/Refractory Multiple myeloma with plasmacytoma Adequate cardiac function , hepatic and renal function Adequate hematopoietic function i. White blood cells ≥3000 ii. Absolute neutrophil count ≥1500 iii. Platelets ≥50,000 iv. Hemoglobin >7.5mg/dL ( Transfusion is not permitted within 2 weeks.) v. Total bilirubin <1.5 times upper limit of normal vi. AST and ALT <1.5 times upper limit of normal vii. Serum creatinine <1.5 times upper limit of normal Singed and dated informed consent of document indicating that the patient(or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment For women of child bearing age, it should be confirmed that they are not pregnant and that they should be contraception during the study period and for up to 3 months after the end of study Male should agree to the barrier method during the study period and up to 3 months after the end of the study

Exclusion Criteria:

* HSCT (hematopoietic stem cell transplantation) within the last 12 weeks
* Other severe acute or

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-12-21 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Complete response rate in terms of plasmacytoma | within 4 weeks after the 3 cycles of combination therapy (daratumumab plus DCEP)
  disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow

SECONDARY OUTCOMES:
Response rate (Complete response + Partial Response) by IMWG criteria | within 4 weeks after the 3 cycles of combination therapy (daratumumab plus DCEP)
  Complete response rate in terms of plasmacytoma plus partial response rate by IMWG criteria
CR rate by IMWG criteria | within 4 weeks after the 3 cycles of combination therapy (daratumumab plus DCEP)
  Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow
Progression free survival | 3,6,12,24 months after the last administration of daratumuamb
  from the last administration date of daratumumab to the date of disease progression or date from any cause
Overall Survival | 3,6,12,24 months after the last administration of daratumuamb
  from the last administration date of daratumumab to death from any cause
Safety and toxicity profile | 3,6,12,24 months the first administration of daratumumab
  according to CTCAE version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: YOUNGIL KOH, MD., Ph.D, Principal Investigator — Seoul National University Hospital; JEONGOK LEE, MD., Ph.D., Study Director — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
IPD regarding participant demographics, study treatment, response, survival, and adverse events will be shared after publishment of the study results.
Supporting Information: Study Protocol
Time Frame: Time Frame:
  IPD will be shared after the publication of the study results without time limit.
Access Criteria: IPD will be shared only for the research purpose.